CLINICAL TRIAL: NCT04801797
Title: A Phase 2 Randomized Study Comparing Venetoclax and Azacitidine to Induction Chemotherapy for Newly Diagnosed Fit Adults With Acute Myeloid Leukemia
Brief Title: Venetoclax + Azacitidine vs. Induction Chemotherapy in AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-113
Record Dates: First submitted 2021-03-08; First posted 2021-03-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Daunorubicin; venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, phase II randomized clinical trial to compare the therapeutic activity of conventional induction chemotherapy (7+3 regimen or liposomal daunorubicin and cytarabine) (Standard arm) to the combination of venetoclax and azacitidine among fit, traditionally induction-eligible adults with newly diagnosed acute myeloid leukemia (AML).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Conventional Induction) (Experimental): Randomized participants will receive cytarabine and idarubicin [or daunorubicin) per standard of care as follows:
  Induction: cytarabine on days 1-7 and idarubicin (or daunorubicin) on days 1-3 of induction.
  Second Induction (if needed): Cytarabine on days 1-5 and idarubicin (or daunorubicin) on days 1-2 of re-induction.
  Consolidation (if needed): If < 60 years, cytarabine days 1,3,5 of consolidation cycles, and if ≥60 years, cytarabine days 1-5 of consolidation cycles
  Those with secondary or therapy-related AML can receive liposomal daunorubicin and cytarabine (Vyxeos) per standard of care as follows:
  Induction: Liposomal daunorubicin and cytarabine (Vyxeos) on Days 1,3, 5 of induction.
  Second Induction (if needed): Liposomal daunorubicin and cytarabine (Vyxeos) on days 1,3 of re-induction Consolidation (if needed): liposomal daunorubicin and cytarabine (Vyxeos) on days 1,3 of consolidation cycles
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Daunorubicin; Drug: Liposomal daunorubicin and cytarabine
- Investigational (Venetoclax and Azacitidine) (Experimental): Participants will receive azacitidine on days 1-7 and venetoclax daily for up to (3) three 28-day study cycles and evaluated for response or benefit. If benefit/response is achieved, azacitidine on days 1-7 and venetoclax on days 1-28 (or less if deemed necessary per protocol) will be given in repeating 28-day cycles until benefit/response is no longer achieved or until patient proceeds to transplantation.
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Cytarabine — Intravenous infusion
  Other Names: Ara-C; Arabinosylcytosine
  Arms: Standard of Care (Conventional Induction)
Drug: Idarubicin — Intravenous infusion
  Arms: Standard of Care (Conventional Induction)
Drug: Daunorubicin — Intravenous infusion
  Arms: Standard of Care (Conventional Induction)
Drug: Liposomal daunorubicin and cytarabine — Intravenous infusion
  Other Names: Vyxeos
  Arms: Standard of Care (Conventional Induction)
Drug: Venetoclax — Orally by mouth
  Other Names: Venclexta
  Arms: Investigational (Venetoclax and Azacitidine)
Drug: Azacitidine — Intravenous infusion
  Other Names: Vidaza
  Arms: Investigational (Venetoclax and Azacitidine)

SUMMARY:
This research is being done to assess the therapeutic activity of a promising combination (azacitidine and venetoclax) versus conventional cytotoxic chemotherapy in induction-eligible patients with acute myeloid leukemia.

This study involves the following:

* Venetoclax and azacitidine (investigational combination)
* Cytarabine and idarubicin or daunorubicin (per standard of care) or Liposomal daunorubicin and cytarabine (per standard of care)

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II randomized clinical trial to compare the therapeutic activity of conventional induction chemotherapy (7+3 regimen or liposomal daunorubicin and cytarabine) to the combination of venetoclax and azacitidine among fit, traditionally induction-eligible adults with newly diagnosed acute myeloid leukemia (AML).

The U.S. Food and Drug Administration (FDA) has approved the combinations of liposomal daunorubicin and cytarabine as well as cytarabine and idarubicin or daunorubicin as treatment options for acute myeloid leukemia (AML)

The FDA has approved the combination of venetoclax and azacitidine for people with acute myeloid leukemia (AML) that are over the age of 75 or who have comorbidities that preclude intensive induction chemotherapy.

Venetoclax may interact with BCL-2 (a protein that initiates tumor growth, disease progression, and drug resistance) and inhibit BLC-2 which can lead to cancer cell death. Azacitidine may cause cell death in rapidly dividing cells, which may lead to cancer cell death since cancer cells do not grow at a normal rate. Induction Chemotherapy which includes the drugs idarubicin or daunorubicin, cytarabine, and liposomal daunorubicin and cytarabine is the standard of care chemotherapy treatment for someone with acute myeloid leukemia (AML).

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

Participants will receive study treatment for as long as they and their doctor believe they are benefitting from the study drugs. Participants will then be followed for 3 years or until they withdraw their consent to be contacted.

It is expected that about 172 people will take part in this research study.

AbbVie, a biopharmaceutical company, is supporting this research study by providing funding for the study, including one of the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participants must have pathologically confirmed, newly diagnosed acute myeloid leukemia (AML), and characterized by 20% or more blasts in the peripheral blood or bone marrow. The AML may be either:

  * De Novo: AML in patients with no clinical history of prior myelodysplastic syndrome (MDS), myeloproliferative disorder, or exposure to potentially leukemogenic therapies or agents
  * Secondary AML (sAML): refers to an acute leukemic process (1) evolving from known prior myelodysplasia, myeloproliferative disorder, or aplastic anemia with or without treatment or; (2) as a product of previous exposure to a proven leukemogenic chemotherapeutic agent
* Eligible for intensive induction chemotherapy, according to their treating physician
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Left ventricular ejection fraction > 50% as measured by echocardiogram or MUGA scan
* Must not have received systemic prior antineoplastic therapy for treatment for the newly diagnosed AML, including radiation therapy, except hydroxyurea for the purposes of cytoreduction. Patients may also have received all-trans retinoic acid (ATRA) if there is an early suspicion of acute promyelocytic leukemia (APL, M3-AML), although if confirmed to have APL these patients will be excluded from the study.
* Adequate renal function as defined by calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula or measured by 24 hours urine collection).
* Adequate hepatic function per local laboratory reference ranges as follows:

  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0X ULN (unless secondary to leukemia, in which case patient may be eligible after consideration and approval by the Overall PI)
  * Total bilirubin ≤ 2.0 x ULN (unless bilirubin rise is known to be due to Gilbert's syndrome or of non-hepatic origin)
* The effects of venetoclax on the developing human fetus are unknown. For this reason and because other chemotherapeutic agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women should use contraceptives for at least 30 days following the last dose of venetoclax. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Diagnosis of Acute promyelocytic leukemia (APL) or AML with favorable cytogenetics [t(8;21), inv(16), t(16;16)]
* Patients < 60 years old with NPM1-mutated AML:
* Patients with FLT3-mutated AML (TKD or ITD) - see notes below.

  * Institutional FLT3 mutational assays can be used to assess for detection of the mutation.
  * A patient with a FLT3 mutation detected at a level of 5% VAF or less, below that typically detectable on the companion diagnostics approved for use by the FDA (http://www.fda.gov/CompanionDiagnostics), would be deemed eligible to enroll.
  * A negative FLT3 mutation result using an outside laboratory assay that is equivalent or similar to that approved as a companion diagnostic by the FDA (http://www.fda.gov/CompanionDiagnostics) is sufficient to rule out FLT3 mutated disease.
* Patients with a known diagnosis of CML or known presence of BCR-Abl alteration
* Patients with acute leukemia with ambiguous lineage or mixed phenotype
* Patients that have received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
* Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Patients who have had prior systemic cytotoxic chemotherapy or radiotherapy for AML (excluding patients with therapy-related AML), except for hydroxyurea or 6-MP as noted. Empiric intrathecal chemotherapy during a diagnostic lumbar puncture is allowed, as long as CNS disease is not suspected.
* Patients treated with prior hypomethylating therapy (such as azacitidine or decitabine).
* Patients who will exceed a lifetime anthracycline exposure of >550 mg/m2 daunorubicin or equivalent (or >400 mg/m2 daunorubicin or equivalent in the event of prior mediastinal radiation) if they receive the maximum potential exposure to anthracyclines per protocol (including both induction and consolidation cycles).
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with a history of other malignancies within 3 years and without any evidence of disease progression may be considered, but only after consideration and approval by the Overall PI. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, breast DCIS, and basal cell or squamous cell carcinoma of the skin.
* Current clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukemic CNS involvement (no lumbar puncture required, clinical assessment per investigator's judgment is sufficient).
* Prior bone marrow transplantation for a myeloid malignancy
* Participants who are receiving any other investigational agents within the prior 14 days.
* Currently clinically active hepatitis C or hepatitis B infection, as suggested by serology or viral load.
* Human immunodeficiency virus (HIV)-infected participants. Patients with detectable viral load on a stable anti-viral regimen may be eligible, after discussion with the study overall PI.
* Current or history of congestive heart failure New York Heart Association (NYHA) class 3 or 4, or any known history of an LVEF <50%, as measured by MUGA scan or echocardiogram. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Known hypersensitivity to the trial drugs or other contraindication to standard "7+3" induction chemotherapy.
* WBC > 25 x 109/L. Note: hydroxyurea is permitted to meet this criterion. If WBC cannot be controlled to <25 x 109/L at the time of enrollment, the WBC management plan must be discussed and approved by the Overall PI.
* Patients who might refuse to receive blood products and/or have a hypersensitivity to blood products
* Patients with clinically significant persistent electrolyte abnormalities such as hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypomagnesemia, and hypermagnesemia of Grade > 1 per NCI CTCAE, v5.0. Treatment for correction of above electrolyte imbalances is permitted during screening to meet eligibility.
* Uncontrolled intercurrent illness including, but not limited to, clinically ongoing or active infection requiring intravenous antibiotics (IV antibiotics are allowed if infection is deemed to be controlled), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known GI disease or GI procedures that could interfere with the oral absorption or tolerance of the study drugs. Examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease.
* Pregnant women are excluded from this study because venetoclax and azacitidine, along with standard induction chemotherapy, carries the potential for teratogenic or abortifacient effects. Because there is potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax as well as azacitidine, cytarabine, daunorubicin and idarubicin, breastfeeding should be avoided. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
* Patients who are otherwise felt unable to comply with the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | From the time from randomization to time for up to 3 years, per protocol.
  Primary endpoint is event-free-survival of patients treated with venetoclax and azacitidine compared to patients treated with standard induction with either 7+3 regimen or liposomal daunorubicin and cytarabine
  Events are described in the protocol and will include
  * Progressive Disease as defined above
  * Any change in therapy due to leukemic persistence.
  * Transition to hospice
  * Relapse following CR, CRi, or CRh
  * Any death
  Assessments of differences in EFS between the randomized arms will be made with the log-rank test; modeling will employ the Cox proportional hazards model. We also plan to assess the difference in estimated EFS at one year, using Kaplan-Meier estimates with standard deviation calculated by Greenwood's formula.
  EFS will be assessed using the Kaplan-Meier method. EFS will be assessed with the log-rank test, and cox proportional hazards model when appropriate.

SECONDARY OUTCOMES:
Rate of response | From the time from randomization to time for up to 6 months.
  Evaluated overall and separately for patients with primary and secondary AML, comparisons will be based on the Fisher exact test.
  CR and CRi will be assessed. Study also includes CRh as a possible response, CRh aims to describe marrow blast clearance and evidence of partial hematologic recovery not captured by current CR or CRi, criteria.
Treatment-related toxicity | Enrollment to end of treatment duration for up to 12 months.
  Assessed using CTCAE 5
Rate of Minimal Residual Disease (MRD) negativity | From time of enrollment until up to the first 6 months.
  Assessed by flow cytometry and next-generation sequencing
30-day mortality | From the time of start of therapy until through the first 30 days.
  Analyzed using the Kaplan Meier method.
60-day mortality | From the time of start of therapy until through the first 60 days.
  Analyzed using the Kaplan Meier method.
Overall survival (OS) | Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive, or for up to 3 years.
  Survival will be summarized using the method of Kaplan Meier, and assessed using the log rank test and Cox proportional hazards when appropriate.
Rate of stem cell transplantation (SCT) following induction | From time of enrollment until up to 3 years following start of treatment.
  The proportion of patients that receive a hematopoietic stem cell transplant following induction therapy or consolidation/continuation therapy.
Patient reported quality of life (QOL) | up to one year
  To compare quality of life between the two groups using the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leuk). the FACT-Leukemia ranges from 0-176 with higher scores indicating better quality of life
Patient-reported depression symptoms | up to one year
  To compare depression symptoms between the two groups using the Hospital Anxiety and Depression Scale (HADS-Depression). the HADS-depression ranges from 0 (no distress) to 21 (maximum distress) with higher scores indicating worse depression symptoms
Patient-reported anxiety symptoms | up to one year
  To compare anxiety symptoms between the two groups using the Hospital Anxieyt and Depression Scale (HADS-Anxiety). the HADS-Anxiety ranges from 0 (no distress) to 21 (maximum distress) with higher scores indicating worse anxiety symptoms
Patient-reported symptom burden | up to one year
  To compare symptom burden between the two groups using the Edmonton Symptom Assessment Scale (ESAS-revised). ESAS ranges from 0-100 with higher scores indicating worse symptom burden
Patient-reported post-traumatic stress symptoms | up to one year
  To compare post-traumatic stress (PTSD) symptoms between the two groups using the PTSD-Checklist-Civilian Version. The PTSD-Checklist ranges from 17-85 with higher scores indicating worse PTSD symptoms
Health care utilization - hospitalizations | up to 1 year
  To compare number of hospitalizations between the two groups using linear regression (and adjusting for any potential imbalances between the groups
Health care utilization - days alive and out of the hospital | up to 1 year
  To compare days alive and out of the hospital between the two groups using linear regression (and adjusting for any potential imbalances between the groups)
Health care utilization - Intensive care unit admissions | up to 1 year
  To compare intensive care unit admissions (yes vs. no) between the two groups using logistic regression (and adjusting for any potential imbalances between the groups)
Cost of care | up to 1 year
  To compare cost of care between the two groups using parametric and non-parametric tests based on distribution of the data
Incidence of neutropenic infections | Up to 8 weeks
  Number of patients that experience neutropenic fever during induction cycles (up to 2 cycles).
100-Day post-transplant mortality | From date of transplantation through 100 days following transplantation.
  Assessed using the Kaplan Meier method
Incidence of grade 3 or greater acute graft versus host disease (GVHD) | Patients that receive a SCT will be followed post-SCT through up to 100 days.
  Assessed among patients that receive HSCT following induction.

CONTACTS AND LOCATIONS:
Overall Officials: Amir T Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - University of California - Davis, Sacramento, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Waclawiczek A, Leppa AM, Renders S, Stumpf K, Reyneri C, Betz B, Janssen M, Shahswar R, Donato E, Karpova D, Thiel V, Unglaub JM, Grabowski S, Gryzik S, Vierbaum L, Schlenk RF, Rollig C, Hundemer M, Pabst C, Heuser M, Raffel S, Muller-Tidow C, Sauer T, Trumpp A. Combinatorial BCL2 Family Expression in Acute Myeloid Leukemia Stem Cells Predicts Clinical Response to Azacitidine/Venetoclax. Cancer Discov. 2023 Jun 2;13(6):1408-1427. doi: 10.1158/2159-8290.CD-22-0939. PMID 36892565